CLINICAL TRIAL: NCT00479947
Title: A Double-Blind,Randomized Placebo-Controlled Study Using Probiotic Lactobacillus GR-1 and RC-14 as an Adjunctive Therapy to Fluconazole in the Treatment of Yeast Vaginitis
Brief Title: Use of Oral Probiotics as an Adjunctive Therapy to Fluconazole in the Treatment of Yeast Vaginitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faith Mediplex (Other)
Collaborators: UrexBiotech (Unknown); Chr Hansen (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UB-CHr-N
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Vaginal Candidiasis
Keywords: Yeast vaginitis; Probiotics; Lactobacilli; Fluconazole
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Probiotics; Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Probiotics (Natural product)
Drug: Probiotics (L. rhamnosus GR-1 and L. reuteri RC-14)

SUMMARY:
Yeast vaginitis is a very common ailment affecting premenopausal women in Nigeria. This condition is more prevalent in the age group between 21-30 years. More than 75% of premenopausal women and university students are diagnosed with yeast infections annually. In most of these women, recurrent rate of vaginal candidiasis with empiric therapy, stands between 70 and 80%. In addition, resistance to anti-fungal agents is increasing at an alarming speed, particularly with species other than Candida albicans such as C tropicalis and C glabrata. The healthy vaginal environment is composed mainly of lactobacilli and when these organisms are suppressed overgrowth of a large number of pathogens occur including yeasts. In this pilot study,we hypothesize that oral administration of two well documented strains of lactobacilli (L.rhamnosis GR-1 and L.reuteri RC-14 ) given to women with recurrent yeast vaginitis, following standard therapy with fluconazole will result in a significant reduction in recurrence rate of the disease.

DETAILED DESCRIPTION:
STUDY HYPOTHESIS The administration of two well documented strains of lactobacilli (L.rhamnosis GR-1 and L.reuteri RC-14 ) given to women with recurrent yeast vaginitis, following standard therapy with fluconazole and compared with placebo will result in a significant reduction in recurrence rate of the disease.

Methodology

Study participants

Inclusion criteria:

* Premenopausal women suffering from acute or chronic yeast vaginitis and a past history of 3 or 4 episodes over the 12 months will be selected.
* All participants must be symptomatic, i.e. the participant must have identified herself as suffering from one or more of the following: abnormal/odourless vaginal discharge, dyspareunia or dysuria, localized irritation or discomfort around the vagina.

Exclusion criteria:

* Participants must not be suffering from other urogenital infections or conditions such as HIV that will potentially alter their response to disease. Participants will be tested and excluded for the presence of Trichomonas vaginalis and Bacterial vaginosis at inclusion. Other conditions will be ruled out on the basis of medical history and clinical assessment.
* Participants must not be pregnant.
* Participants must not be younger than 18 or older than 50 years.
* Participants must not be menstruating during diagnosis or treatment

Laboratory Diagnosis:

Microscopic examination of vaginal secretion in 10% KOH for hyphae and mycelia Culture for fungal agent using Sabbraoud agar/broth.

Randomisation:

• Participants randomised for age, history of previous (past year) yeast vaginitis.

Treatment Protocol 100 premenopausal women presenting with acute yeast vaginitis and a past history of 3 or 4 episodes of yeast vaginitis over the past 12 months will be treated with one oral dose of Fluconazole (Diflucan), then randomized into 2 groups:

* Group A: Receiving one oral dose of Fluconazole + oral placebo capsules for 3 months.
* Group B: Receiving one oral dose of Fluconazole + capsules of L. rhamnosus GR-1 and L reuteri RC-14 containing 5 billion live organisms for 3 months.

Both groups of patients will be followed at 7days for proof of cure, 1 month, 2 months and 3 months following enrolment.

At all follow-up visits, the patients will be checked for symptoms and examined physically. Vaginal swabs will be tested for fungi microscopically and by culture, and BV organisms using Nugent scoring or with BV Blue test kit for vaginal sialidase.

Data to be collected

Symptoms:

* Lifestyle questionnaire, to include daily self-assessment of presence and severity of condition (discharge, irritation,) for the first 7 days. To include self-determined definition of when recovery begins and when it is complete. Also include menstrual cycle information (during the treatment, is the subject in early, mid or late cycle?).
* Physician assessment at each visit.

Vaginal swabs - two per visit:

* Day 0 (before treatment)
* Day 7 (Proof of cure for the two groups).

  * 1 month after treatment
  * 2 months after treatment
  * 3 months after treatment.

Statistical Analysis

In the placebo group of patients, it is anticipated that at the 3 month period, a recurrence rate of 50% will occur, whereas, in the treatment arm a reduction in recurrence to 25% will be achieved. The study is designed to have a power of 80% and to detect a reduction in recurrence at two-sided 5% significance level.

Participants Recruitment:

Subjects will be recruited from the women attending urogenital tract infection clinics at Faith Mediplex, Benin City.

Risk No risks are expected except the usual adverse effects associated with Fluconazole, otherwise probiotic lactobacilli are generally regarded as safe (GRAS) and no known side effects have been attributed to probiotic lactobacilli in immunocompetent individuals.

Benefits There may be benefits accruing from the probiotic arm of the study as recurrence rate may be low than the placebo. Also there may not be any direct benefit, but information gathered will help us in evaluating whether oral use of probiotics could be practically applicable in our environment against vaginal yeast infections.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women suffering from acute or chronic yeast vaginitis and a past history of 3 or 4 episodes over the 12 months will be selected.
* All participants must be symptomatic, i.e. the participant must have identified herself as suffering from one or more of the following: abnormal/odourless vaginal discharge, dyspareunia or dysuria, localized irritation or discomfort around the vagina.

Exclusion Criteria:

* Participants must not be suffering from other urogenital infections or conditions such as HIV that will potentially alter their response to disease. Participants will be tested and excluded for the presence of Trichomonas vaginalis and Bacterial vaginosis at inclusion. Other conditions will be ruled out on the basis of medical history and clinical assessment.
* Participants must not be pregnant.
* Participants must not be younger than 18 or older than 50 years.
* Participants must not be menstruating during diagnosis or treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
In the placebo group of patients, it is anticipated that at the 3 month period, a recurrence rate of 50% will occur, whereas, in the treatment arm a reduction in recurrence to 25% will be achieved | 3 months

SECONDARY OUTCOMES:
Reduction in clinic visits for urogenital care and cost savings | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chinonye C EZE-OKOROIKPA, MBBS, Study Chair — Faith Mediplex; MARTIN U DURU, MSc, Study Director — Faith Mediplex; KINGSLEY C ANUKAM, PhD, Principal Investigator — Benson Idahosa University, Benin City and Canadian R & D Centre for Probiotics, Lawson Health Research Intsitute, London, Ontario, Canada. anukamkc@yahoo.com; ALFRED AIYEBELEHIN, MBBS, Study Chair — Faith Mediplex
Locations (1):
- FaithMediplex, Benin City, Edo, Nigeria

REFERENCES:
- [Background] Falagas ME, Betsi GI, Athanasiou S. Probiotics for prevention of recurrent vulvovaginal candidiasis: a review. J Antimicrob Chemother. 2006 Aug;58(2):266-72. doi: 10.1093/jac/dkl246. Epub 2006 Jun 21. PMID 16790461
- [Background] Osset J, Garcia E, Bartolome RM, Andreu A. [Role of Lactobacillus as protector against vaginal candidiasis]. Med Clin (Barc). 2001 Sep 22;117(8):285-8. doi: 10.1016/s0025-7753(01)72089-1. Spanish. PMID 11571120